CLINICAL TRIAL: NCT07036003
Title: Recombinant Human Growth Hormone (rHGH) for Knee Osteoarthritis (KORR): a Pilot, Randomized Placebo-controlled Trial
Brief Title: Recombinant Human Growth Hormone (rHGH) for Knee Osteoarthritis (KORR)
Acronym: KORR
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dr. David Wasserstein (Other)
Collaborators: Sunnybrook Research Institute (Other)
Responsible Party: Sponsor-Investigator, Dr. David Wasserstein, Assistant Professor - University of Toronto; Associate Scientist - Sunnybrook Research Institute, Sunnybrook Health Sciences Centre
Organization: Sunnybrook Health Sciences Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6427
Record Dates: First submitted 2025-05-30; First posted 2025-06-25 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis (Knee OA); Knee Osteoarthritis (OA)
Keywords: Recombinant Human Growth Hormone; rHGH; Saizen; Knee Osteoarthritis; Knee OA
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Recombinant Human Growth Hormone (rHGH) (Experimental): Self-administered subcutaneous injection into the abdomen or gluteal region once per day for six weeks.
  Interventions: Drug: Somatropin (recombinant human growth hormone)
- Bacteriostatic Saline (Placebo Comparator): Self-administered subcutaneous injection into the abdomen or gluteal region once per day for six weeks.
  Interventions: Drug: bacteriostatic saline placebo

INTERVENTIONS:
Drug: Somatropin (recombinant human growth hormone) — Study participants will deliver Somatropin via self-administered subcutaneous injection into the abdomen or gluteal region once per day for six weeks at a dose of 0.5mg/day per body surface area (0.5mg/m2/day).
  Arms: Recombinant Human Growth Hormone (rHGH)
Drug: bacteriostatic saline placebo — Study participants will deliver bacteriostatic saline via self-administered subcutaneous injection into the abdomen or gluteal region once per day for six weeks in an identical delivery device to the experimental arm.
  Arms: Bacteriostatic Saline

SUMMARY:
The goal of this clinical trial is to see if people with knee osteoarthritis would be willing to comply and adhere to incorporating Recombinant Human Growth Hormone (rHGH), specifically Saizen Somatropin solution, into their treatment plan.

Participants will be asked to:

* Self-inject the treatment solution (placebo or somatropin) into the abdominal or gluteal area once per day for a total of 6 weeks.
* Complete questionnaires related to their knee pain and activities of daily living.
* Provide blood tests.
* Complete various measurements including: circumference of thigh, calf, and abdomen; strength of thigh and knee; range of motion of both knees; and gait analysis.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 - 60 years old.
* Diagnosis of isolated knee osteoarthritis for greater than 6 months.

Exclusion Criteria:

* Previous or pending surgery to involved knee.
* Previous major trauma to involved knee, or ipsilateral knee, hip, or ankle.
* Recent (less than 6 months) intra-articular injection into the involved knee.
* High grade ligamentous knee injury.
* Known allergy to recombinant human growth hormone (rHGH) or reconstitutive solutions.
* BMI of less than 20 or greater than 35.
* Documented history of growth disorder of bones or connective tissue, type 1 or 2 diabetes, myopathy, cancer, endocrine disorder, severe hypertension (SBP > 180) or rheumatologic disorder.
* Pregnant or breastfeeding, or actively attempting to get pregnant.
* Currently on hypoglycemic therapy, oral estrogen or glucocorticoid replacement therapy.
* Would have difficulty with the self-injection schedule or other cognitive/ functional limitations.
* Vital signs or routine bloodwork outside of normal range.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the medication administration | 6 weeks after treatment begins.
  Participant adheres to self-administration of injections once daily for 6 weeks.

SECONDARY OUTCOMES:
Clinical Outcomes: knee extension strength | At 6 weeks and 24 months time points after enrolment
  Participants' knee extension strength will be measured using HUMAC Norm Extremity Strength Testing system.
Clinical Outcome: knee flexion strength | At 24 months after enrolment.
  Participants' knee flexion strength will be measured using HUMAC Norm Extremity Strength Testing system.
Clinical Outcomes: thigh muscle strength | At baseline, 6 weeks, 3 months, 6 months, 12 months, and 24 months study visits.
  Participants' thigh muscle strength will be measured through hip flexion, hip abduction and knee flexion using a goniometer.
Clinical Outcomes: Kinematic Gait Analysis | At baseline, 6 weeks and 6 months study visits.
  Participants' kinematic gait analysis will be measured with single/ two leg hop/jump and single/ two leg squat, using the Theia Markerless system before and after treatment.
Thigh circumference | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participant's measurements of function will be measured by their thigh circumference compared to the contralateral leg, and baseline.
Mid-calf circumference | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participant's measurements of function will be measured by their mid-calf circumference compared to the contralateral leg, and baseline.
Abdominal circumference | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participant's measurements of function will be measured by their abdominal circumference.
Range of motion of both knees | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participant's measurements of function will be measured by Range of motion of both knees.
6 Minute Walk Test (6MWT) | At baseline, 6 weeks, 3 months, 6 months, and 12 months after enrolment.
  Participants' distance traveled in the span of 6 minutes will be measured on a treadmill (unit: total meters).
Activity Count | From enrolment to the 12-week study visit.
  Participants' activity count will be measured using a fitness tracker (ActiGraph) worn around the ankle. The total time the fitness tracker is worn will be monitored by the device.
Knee Injury and Osteoarthritis Score (KOOS) | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participants will be asked to complete the Knee Injury and Osteoarthritis Score (KOOS) questionnaire to measure their overall well-being.
  KOOS uses a Likert scale ranging from 0 (No problems) to 4 (Extreme problems).
20-Item Short Form Survey (SF-20) | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participants will be asked to complete the 20-Item Short Form Survey Instrument (SF-20) questionnaire which measures their overall well-being including their physical and social functioning.
Tegner Activity Scale | At baseline, 6 weeks, 3, 6, 12 and 24 months study visits
  Participants will be asked to complete the Tegner Activity Scale questionnaire, which measures their level of activity.
  A 11-point scale (ranging from 0 - 10) is used where a higher score indicates higher level of activity.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Wasserstein, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Statement: All data relevant to the study will be included in the final study manuscript or uploaded as supplementary information.
  Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be able to access the IPD and supporting information to achieve aims in the approved proposal.
  Proposals should be directed to david.wasserstein@sunnybrook.ca. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Barake M, Klibanski A, Tritos NA. Effects of recombinant human growth hormone therapy on bone mineral density in adults with growth hormone deficiency: a meta-analysis. J Clin Endocrinol Metab. 2014 Mar;99(3):852-60. doi: 10.1210/jc.2013-3921. Epub 2014 Jan 1. PMID 24423364
- [Background] Yeo AL, Levy D, Martin FC, Sonksen P, Sturgess I, Wheeler MM, Young A. Frailty and the biochemical effects of recombinant human growth hormone in women after surgery for hip fracture. Growth Horm IGF Res. 2003 Dec;13(6):361-70. doi: 10.1016/j.ghir.2003.08.001. PMID 14624771
- [Background] Tavares AB, Micmacher E, Biesek S, Assumpcao R, Redorat R, Veloso U, Vaisman M, Farinatti PT, Conceicao F. Effects of Growth Hormone Administration on Muscle Strength in Men over 50 Years Old. Int J Endocrinol. 2013;2013:942030. doi: 10.1155/2013/942030. Epub 2013 Dec 8. PMID 24382963
- [Background] Rahimzadeh P, Imani F, Faiz SH, Alebouyeh MR, Azad-Ehyaei D, Bahari L, Memarian A, Kim KH. Adding Intra-Articular Growth Hormone to Platelet Rich Plasma under Ultrasound Guidance in Knee Osteoarthritis: A Comparative Double-Blind Clinical Trial. Anesth Pain Med. 2016 Oct 19;6(6):e41719. doi: 10.5812/aapm.41719. eCollection 2016 Dec. PMID 28975078
- [Background] Dunn AR. Intra-articular growth hormone injections regrow cartilage, increase motion and reduce pain in 93 per cent. of arthritic ankles. Osteoarthritis Cartilage. 2012;20:S295-S296. doi:10.1016/j.joca.2012.02.512
- [Background] Yang S, Cao L, Cai S, Yuan J, Wang J. A systematic review of growth hormone for hip fractures. Growth Horm IGF Res. 2012 Jun-Aug;22(3-4):97-101. doi: 10.1016/j.ghir.2012.03.002. Epub 2012 Apr 1. PMID 22472350
- [Background] Yarasheski KE, Campbell JA, Smith K, Rennie MJ, Holloszy JO, Bier DM. Effect of growth hormone and resistance exercise on muscle growth in young men. Am J Physiol. 1992 Mar;262(3 Pt 1):E261-7. doi: 10.1152/ajpendo.1992.262.3.E261. PMID 1550219
- [Background] Dubiel R, Callender L, Dunklin C, Harper C, Bennett M, Kreber L, Auchus R, Diaz-Arrastia R. Phase 2 Randomized, Placebo-Controlled Clinical Trial of Recombinant Human Growth Hormone (rhGH) During Rehabilitation From Traumatic Brain Injury. Front Endocrinol (Lausanne). 2018 Sep 10;9:520. doi: 10.3389/fendo.2018.00520. eCollection 2018. PMID 30250451
- [Background] Abreu ME, Valiati R, Hubler R, Moraes AN, Antonini F, de Oliveira Hdo C, Pagnoncelli RM. Effect of Recombinant Human Growth Hormone on Osseointegration of Titanium Implants: A Histologic and Biomechanical Study in Rabbits. J Oral Implantol. 2015 Aug;41(4):e102-9. doi: 10.1563/aaid-joi-D-13-00306. Epub 2014 Jun 19. PMID 24946138
- [Background] Ehrnberg A, Brosjo O, Laftman P, Nilsson O, Stromberg L. Enhancement of bone formation in rabbits by recombinant human growth hormone. Acta Orthop Scand. 1993 Oct;64(5):562-6. doi: 10.3109/17453679308993693. PMID 8237325
- [Background] Raschke MJ, Bail H, Windhagen HJ, Kolbeck SF, Weiler A, Raun K, Kappelgard A, Skiaerbaek C, Haas NP. Recombinant growth hormone accelerates bone regenerate consolidation in distraction osteogenesis. Bone. 1999 Feb;24(2):81-8. doi: 10.1016/s8756-3282(98)00158-6. PMID 9951774
- [Background] Kim SB, Kwon DR, Kwak H, Shin YB, Han HJ, Lee JH, Choi SH. Additive effects of intra-articular injection of growth hormone and hyaluronic acid in rabbit model of collagenase-induced osteoarthritis. J Korean Med Sci. 2010 May;25(5):776-80. doi: 10.3346/jkms.2010.25.5.776. Epub 2010 Apr 16. PMID 20436717
- [Background] Hao Y, Dai K, Guo L, Wang Y, Tang T. Effects of recombinant human growth hormone (r-hGH) on experimental osteoporotic fracture healing. Chin J Traumatol. 2001 May;4(2):102-5. PMID 11834155
- [Background] Lubis AMT, Wijaya MT, Priosoeryanto BP, Saleh RF, Farqani S. Comparison of weekly and single dose intraarticular recombinant human growth hormone injection on cartilage degeneration in osteoarthritic model of white New Zealand rabbits. J Exp Orthop. 2022 Feb 21;9(1):19. doi: 10.1186/s40634-022-00458-y. No abstract available. PMID 35190919
- [Background] Lubis AMT, Wonggokusuma E, Marsetio AF. Intra-articular Recombinant Human Growth Hormone Injection Compared with Hyaluronic Acid and Placebo for an Osteoarthritis Model of New Zealand Rabbits. Knee Surg Relat Res. 2019 Mar 1;31(1):44-53. doi: 10.5792/ksrr.18.062. PMID 30871292
- [Background] Boesen AP, Dideriksen K, Couppe C, Magnusson SP, Schjerling P, Boesen M, Kjaer M, Langberg H. Tendon and skeletal muscle matrix gene expression and functional responses to immobilisation and rehabilitation in young males: effect of growth hormone administration. J Physiol. 2013 Dec 1;591(23):6039-52. doi: 10.1113/jphysiol.2013.261263. Epub 2013 Sep 30. PMID 24081158
- [Background] Linderman JK, Gosselink KL, Booth FW, Mukku VR, Grindeland RE. Resistance exercise and growth hormone as countermeasures for skeletal muscle atrophy in hindlimb-suspended rats. Am J Physiol. 1994 Aug;267(2 Pt 2):R365-71. doi: 10.1152/ajpregu.1994.267.2.R365. PMID 8067444
- [Background] Dalla Libera L, Ravara B, Volterrani M, Gobbo V, Della Barbera M, Angelini A, Danieli Betto D, Germinario E, Vescovo G. Beneficial effects of GH/IGF-1 on skeletal muscle atrophy and function in experimental heart failure. Am J Physiol Cell Physiol. 2004 Jan;286(1):C138-44. doi: 10.1152/ajpcell.00114.2003. Epub 2003 Sep 17. PMID 13679302
- [Background] Newman CB, Carmichael JD, Kleinberg DL. Effects of low dose versus high dose human growth hormone on body composition and lipids in adults with GH deficiency: a meta-analysis of placebo-controlled randomized trials. Pituitary. 2015 Jun;18(3):297-305. doi: 10.1007/s11102-014-0571-z. PMID 24810900
- [Background] Vinciguerra M, Musaro A, Rosenthal N. Regulation of muscle atrophy in aging and disease. Adv Exp Med Biol. 2010;694:211-33. doi: 10.1007/978-1-4419-7002-2_15. PMID 20886766
- [Background] Favier FB, Benoit H, Freyssenet D. Cellular and molecular events controlling skeletal muscle mass in response to altered use. Pflugers Arch. 2008 Jun;456(3):587-600. doi: 10.1007/s00424-007-0423-z. Epub 2008 Jan 12. PMID 18193272
- [Background] Al-Samerria S, Radovick S. The Role of Insulin-like Growth Factor-1 (IGF-1) in the Control of Neuroendocrine Regulation of Growth. Cells. 2021 Oct 5;10(10):2664. doi: 10.3390/cells10102664. PMID 34685644
- [Background] Brinkman JE, Tariq MA, Leavitt L, Sharma S. Physiology, Growth Hormone. 2023 May 1. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK482141/ PMID 29489209
- [Background] Hoglund LT, Pontiggia L, Kelly JD 4th. A 6-week hip muscle strengthening and lumbopelvic-hip core stabilization program to improve pain, function, and quality of life in persons with patellofemoral osteoarthritis: a feasibility pilot study. Pilot Feasibility Stud. 2018 Apr 6;4:70. doi: 10.1186/s40814-018-0262-z. eCollection 2018. PMID 29636983
- [Background] Brosseau L, Taki J, Desjardins B, Thevenot O, Fransen M, Wells GA, Mizusaki Imoto A, Toupin-April K, Westby M, Alvarez Gallardo IC, Gifford W, Laferriere L, Rahman P, Loew L, De Angelis G, Cavallo S, Shallwani SM, Aburub A, Bennell KL, Van der Esch M, Simic M, McConnell S, Harmer A, Kenny GP, Paterson G, Regnaux JP, Lefevre-Colau MM, McLean L. The Ottawa panel clinical practice guidelines for the management of knee osteoarthritis. Part two: strengthening exercise programs. Clin Rehabil. 2017 May;31(5):596-611. doi: 10.1177/0269215517691084. Epub 2017 Feb 1. PMID 28183213
- [Background] Brosseau L, Taki J, Desjardins B, Thevenot O, Fransen M, Wells GA, Mizusaki Imoto A, Toupin-April K, Westby M, Alvarez Gallardo IC, Gifford W, Laferriere L, Rahman P, Loew L, De Angelis G, Cavallo S, Shallwani SM, Aburub A, Bennell KL, Van der Esch M, Simic M, McConnell S, Harmer A, Kenny GP, Paterson G, Regnaux JP, Lefevre-Colau MM, McLean L. The Ottawa panel clinical practice guidelines for the management of knee osteoarthritis. Part three: aerobic exercise programs. Clin Rehabil. 2017 May;31(5):612-624. doi: 10.1177/0269215517691085. Epub 2017 Feb 9. PMID 28183194
- [Background] Brosseau L, Taki J, McLean L. The Ottawa panel clinical practice guidelines for the management of knee osteoarthritis. Part one: introduction, and mind-body exercise programs. Accessed October 15, 2024. https://journals-sagepub- com.myaccess.library.utoronto.ca/doi/10.1177/0269215517691083?icid=int.sj-full- text.similar-articles.2
- [Background] Segal NA, Glass NA, Felson DT, Hurley M, Yang M, Nevitt M, Lewis CE, Torner JC. Effect of quadriceps strength and proprioception on risk for knee osteoarthritis. Med Sci Sports Exerc. 2010 Nov;42(11):2081-8. doi: 10.1249/MSS.0b013e3181dd902e. PMID 20351594
- [Background] Lewek MD, Rudolph KS, Snyder-Mackler L. Quadriceps femoris muscle weakness and activation failure in patients with symptomatic knee osteoarthritis. J Orthop Res. 2004 Jan;22(1):110-5. doi: 10.1016/S0736-0266(03)00154-2. PMID 14656668
- [Background] Amoako AO, Pujalte GG. Osteoarthritis in young, active, and athletic individuals. Clin Med Insights Arthritis Musculoskelet Disord. 2014 May 22;7:27-32. doi: 10.4137/CMAMD.S14386. eCollection 2014. PMID 24899825
- [Background] Khan M, Adili A, Winemaker M, Bhandari M. Management of osteoarthritis of the knee in younger patients. CMAJ. 2018 Jan 22;190(3):E72-E79. doi: 10.1503/cmaj.170696. No abstract available. PMID 29358201
- [Background] Li CS, Karlsson J, Winemaker M, Sancheti P, Bhandari M. Orthopedic surgeons feel that there is a treatment gap in management of early OA: international survey. Knee Surg Sports Traumatol Arthrosc. 2014 Feb;22(2):363-78. doi: 10.1007/s00167-013-2529-5. Epub 2013 Jun 18. PMID 23775341
- [Background] Mendias CL, Enselman ERS, Olszewski AM, Gumucio JP, Edon DL, Konnaris MA, Carpenter JE, Awan TM, Jacobson JA, Gagnier JJ, Barkan AL, Bedi A. The Use of Recombinant Human Growth Hormone to Protect Against Muscle Weakness in Patients Undergoing Anterior Cruciate Ligament Reconstruction: A Pilot, Randomized Placebo-Controlled Trial. Am J Sports Med. 2020 Jul;48(8):1916-1928. doi: 10.1177/0363546520920591. Epub 2020 May 26. PMID 32452208
- [Background] Brophy RH, Fillingham YA. AAOS Clinical Practice Guideline Summary: Management of Osteoarthritis of the Knee (Nonarthroplasty), Third Edition. J Am Acad Orthop Surg. 2022 May 1;30(9):e721-e729. doi: 10.5435/JAAOS-D-21-01233. PMID 35383651
- [Derived] Shah A, Ravi B, Tomescu S, Catapano M, Burkhart TA, Whyne C, Kiss A, Marks P, Wasserstein DN. Recombinant human growth hormone (rHGH) for muscle enhancement in knee osteoarthritis: protocol for a pilot, randomised placebo-controlled trial. BMJ Open. 2026 Feb 4;16(2):e106999. doi: 10.1136/bmjopen-2025-106999. PMID 41638751
- See also: Saizen Drug Monograph. Accessed October 15, 2024. — https://www.emdserono.com/us-en/pi/saizen-ce-pi.pdf